CLINICAL TRIAL: NCT05653973
Title: Protective Mechanisms of Prenatal Aspirin Therapy on Maternal Vascular Dysfunction Following Preeclampsia
Brief Title: Prenatal Aspirin and Postpartum Vascular Function
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anna Stanhewicz, PhD (Other)
Responsible Party: Sponsor-Investigator, Anna Stanhewicz, PhD, Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 202203433
Record Dates: First submitted 2022-12-07; First posted 2022-12-16 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia; Microvascular Function
MeSH Terms: conditions — Pre-Eclampsia | interventions — Acetylcholine; Endothelin-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- assessment of microvascular function (Experimental): The investigators use intradermal microdialysis to deliver acetylcholine, acetylcholine + L-NAME, endothelin-1, endothelin-1 + BQ-788, and endothelin-1 + BQ-123 to the cutaneous microvasculature.
  Interventions: Drug: Acetylcholine; Drug: Endothelin-1

INTERVENTIONS:
Drug: Acetylcholine — acetylcholine, and acetylcholine + L-NAME (Nitric oxide synthase inhibitor) are locally and acutely delivered to the cutaneous microvasculature to assess endothelium- and nitric oxide-dependent dilation
Drug: Endothelin-1 — endothelin-1, endothelin-1 + BQ-788 (endothelin receptor type B-inhibitor), and endothelin-1 + BQ-123 (endothelin receptor type A-inhibitor) are locally and acutely delivered to the cutaneous microvasculature to assess endothelin-mediated constriction and the role of the receptor subtypes in this response.

SUMMARY:
Preeclampsia is a pregnancy disorder affecting ~5-10% of pregnancies in the United States. Women who develop preeclampsia during pregnancy are more likely to develop and die of cardiovascular disease later in life, even if they are otherwise healthy. The reason why this occurs is unclear but may be related to blood vessel damage and increased inflammation that occurs during the preeclamptic pregnancy and persists postpartum. Low dose aspirin (LDA; 75-150mg/daily) is currently the most effective and clinically accepted therapy for reducing preeclampsia prevalence in women at high risk for developing the syndrome. The purpose of this study is to interrogate the mechanisms by which LDA therapy mitigates persistent vascular dysfunction in postpartum women who have had preeclampsia.

In this study, the investigators use the blood vessels in the skin as a representative vascular bed for examining mechanisms of microvascular dysfunction in humans. Using a minimally invasive technique (intradermal microdialysis for the local delivery of pharmaceutical agents) they examine the blood vessels in a dime-sized area of the skin in women who have had a history of preeclampsia. As a compliment to these measurements, they also draw blood from the subjects and isolate the inflammatory cells.

ELIGIBILITY:
Inclusion:

* 18 years or older,
* 12 weeks to 5 years postpartum
* and one of the following:

  1. women who had a normal pregnancy and did not use low does aspirin (LDA) during pregnancy,
  2. women who had a normal pregnancy and used LDA during pregnancy,
  3. women who had preeclampsia and did not use LDA during pregnancy,
  4. women who had preeclampsia and used LDA during pregnancy.

Exclusion:

* current daily aspirin use,
* skin diseases,
* current tobacco use,
* diagnosed or suspected hepatic or metabolic disease including chronic kidney disease (CKD) defined as reduced eGFR < 60 mL/min/1.73m2,
* statin or other cholesterol-lowering medication,
* current antihypertensive medication,
* history of hypertension prior to pregnancy,
* history of gestational diabetes,
* current pregnancy,
* body mass index <18.5 kg/m2,
* allergy to materials used during the experiment.(e.g. latex),
* known allergies to study drugs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
microvascular endothelial function | at the study visit, an average of 4 hours
  cutaneous vascular vasodilator response to exogenous acetylcholine perfusion; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of acetylcholine alone or co-infused with L-NAME
microvascular endothelin-1-mediated constriction | at the study visit, an average of 4 hours
  cutaneous vascular response to exogenous endothelin-1 perfusion; measured with laser-Doppler flowmetry coupled with intradermal microdialysis delivery of endothelin-1 alone or co-infused with BQ-788 or BQ-123

CONTACTS AND LOCATIONS:
Locations (1):
- University of Iowa, Iowa City, Iowa, United States